CLINICAL TRIAL: NCT03451838
Title: The Prediction of Fetal Macrosomia by Measurement of Placenta Volume and Thickness in Pregnant Women With Diabetes Mellitus
Brief Title: Prediction of Fetal Macrosomia by US
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: macrosomia prediction
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Fetal Macrosomia
MeSH Terms: conditions — Fetal Macrosomia | interventions — Ultrasonography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes mellitus: Pregnant women with diabetes mellitus will be examined by us to measures placental volume and thickness ,IV thickness and HbA1c
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: HbA1c level in blood
- control group: Pregnant women with no medical disorders will be examined by us to measures placental volume and thickness ,IV thickness and HbA1c
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: HbA1c level in blood

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound will be done to every pregnant lady
Diagnostic Test: HbA1c level in blood — a blood sample will be taken to measure HbA1c level

SUMMARY:
Fetal macrosomia defined as birth weight above 90th centile ,macrosomia occurs in 42-62%of pregnancy complicated by type 1 diabetes mellitus ,in 30-56% of pregnancy complicated by type 2 diabetes mellitus .

-The delivery of macrosomic infant has potentially severe consequence for both the newborn and mother .Increased birth weight increase the risk in the fetus of shoulder dystocia and premature brachial plexus injury ,and those infant weighing above 4500g are at increased risk for neonatal morbidity ,including the need for assisted ventilation and meconium aspiration .Maternal complication result from operative delivery and include postpartum hemorrhage ,third or fourth degree laceration and postpartum infection .

DETAILED DESCRIPTION:
Estimated fetal body weight is needed especially when head measurement is impossible whenever the fetal head is positioned low in pelvic brim .A convenient method for estimating fetal body weight without head measurement was thus required .

-The human placenta develop with the principal function of providing nutrients and oxygen to the fetus ,adequate fetal growth and subsequent normal birth weight depend on normal placenta .

ELIGIBILITY:
Inclusion Criteria:

* 1.Singleton gestational 2.Gestational age over 16-20 weeks 3.Intact membrane 4.Normal umbilical morphology (two arteries and one vein )

Exclusion Criteria:

1. The presence of fetal congenital anomaly .
2. Multifetal pregnancy.
3. Maternal chronic disease (hypertension, renal disease ,and pulmonary disease ,etc.)
4. Patient with a diagnosis such as oligohydramnios ,preeclampsia and intrauterine growth retardation .
5. Patient who used cigarette or alcohol during pregnancy.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: Singleton gestational Gestational age over 16-20 weeks with Intact membrane with Normal umbilical morphology (two arteries and one vein ) with DM in one group and no medical disorders in another group
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-05-05 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
the number of paticipants who will have babies with macrosomias | within a week from delivery
  To detect number of fetuses who will develop macrosomia

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt; Ahmed samy, M.D, Study Chair — kasraliny hospital- Aljazeerah hospital
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
the data that willbe obtained from this research will be published